CLINICAL TRIAL: NCT02439723
Title: A Phase I, Open Label Study of the Effects of Lean Body Mass (LBM) and Proton Pump Inhibitors (PPIs) on Pharmacokinetics and Safety of Regorafenib (BAY 73-4506) in Cancer Patients
Brief Title: Effects of LBM and PPIs on Pharmacokinetics and Safety of Regorafenib (BAY 73-4506) in Cancer Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawal of supply of investigational product
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Regorafenib 1.0
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Metastatic Solid Malignancies; Locally Advanced Solid Malignancies
Keywords: Regorafenib; Lean body mass; Proton pump inhibitors pharmacokinetics
MeSH Terms: interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regorafenib (Experimental): All patients will be treated with 160 mg regorafenib taken orally once daily for the first 21 days of each 28-day cycle. Doses are to be taken immediately following a light breakfast. During the seven-day break period of cycle 1, patients will start pantoprazole 40 mg twice daily for 8 days
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: Regorafenib
  Other Names: BAY 73-4506; Stivarga

SUMMARY:
The FDA and Health Canada have approved regorafenib at a daily dose of 160mg for the treatment of metastatic colorectal cancer and gastrointestinal stromal cancer; however, the 160 mg dose is not well tolerated by patients, especially women. The purpose of this study is to determine if lean body mass and acidity in the intestinal tract impact how regorafenib is absorbed into the bloodstream and then broken down and removed from the body. This may explain the side effects experienced at the 160 mg dose, especially by women, and inform regorafenib dosing in the future.

DETAILED DESCRIPTION:
Numerous investigators have noted that the recommended flat dosing of regorafenib of 160 mg orally, once daily is not well tolerated by patients, especially women. The purpose of this study is to determine if there is a correlation between lean body mass and regorafenib pharmacokinetics and if so, then it may be possible to exploit this relationship to better dose regorafenib.

Additionally, Bayer has noted that regorafenib steady state levels were lower in gastrointestinal stromal tumour (GIST) patients than in patients with metastatic colorectal cancer. GIST patients have often had gastrectomies that would lead to an elevated pH in the intestinal tract. If regorafenib has a pH dependent solubility then lower regorafenib levels could be due to reduced acidity. The purpose of the second part of the study is to examine the regorafenib pharmacokinetic profile in patients treated with a proton pump inhibitor (pantoprazole) for 7 days, mimicking the altered intestinal environment seen in GIST patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any study procedures completed.
* Subjects with historically confirmed advanced metastatic or refractory solid malignancy who are not candidates for standard therapy.
* Male/female subjects ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2.
* Women of childbearing potential must have a negative urine pregnancy test performed within 7 days before starting study treatment. Women of childbearing potential and men must agree to use adequate contraception since the signing of informed consent until at least 8 weeks after the last study drug administration.
* Life expectancy of at least 8 weeks.
* Adequate bone marrow, and liver function as assessed by the designated laboratory levels within 7 days of starting study treatment:

  1. Platelet count ≥ 100,000/cubic millimeters, hemoglobin (Hb) ≥ 8.0 g/dl, absolute neutrophil count (ANC) ≥ 1500 cubic millimeters
  2. total bilirubin ≤ 1.5 times the upper limit of normal range (ULN). Mildly elevated total bilirubin (<6 mg/dL) is allowed if Gilbert's syndrome is documented
  3. Alanine aminotransferase (ALT) and asparate aminotransferase (AST) ≤ 2.5 times ULN (≤ 5 times ULN for subjects whose cancer involves their liver including liver metastasis).
  4. Alkaline phosphatase limit ≤ 2.5 times ULN (≤ 5 ULN for subjects whose cancer involves their liver including liver metastasis)
  5. Amylase and lipase ≤ 1.5 times ULN
* International normalized ratio (INR) ≤ 1.5 x ULN and partial thromboplastin time (PTT) ≤ 1.5 times ULN. Subjects who are being treated with heparin or warfarin are allowed to participate.
* Estimated glomerular filtration rate (eGFR) ≥ 60 mL/minute as calculated using the Cockcroft-Gault formula

Exclusion Criteria:

* Prior treatment with regorafenib. Patients permanently withdrawn from the study will not be allowed to re-enter the study
* Symptomatic metastatic brain or meningeal tumors unless the patient is greater than 6 months from definitive therapy, has no evidence of tumor growth on an imaging study within four weeks prior to study entry and is not on dexamethasone and clinically stable with respect to the tumor at the time of surgery.
* Major surgery, open biopsy or significant traumatic injury within 28 days before starting the study treatment.
* History of organ allograft.
* Non-healing wound, skin ulcer or bone fracture.
* Uncontrolled intercurrent medical illness including uncontrolled hypertension defined as systolic blood pressure > 150 millimeters of mercury (mmHg) or diastolic blood pressure > 90 mmHg, despite medical management
* History of cardiac disease: congestive heart failure > New York Heart Association (NYHA) Class II; unstable angina (symptoms of angina at rest), new-onset angina (within the last 3 months), myocardial infarction within the past 6 months prior to screening (Visit 1); cardiac ventricular arrhythmias requiring anti-arrhythmic therapy (expect for beta-blockers and digoxin).
* Pleural effusion or ascites with causes respiratory compromise (National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 Grade ≥ 2 dyspnea).
* Interstitial lung disease with ongoing signs and symptoms within 28 days before starting the study treatment
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before the start of study medication.
* Subjects with evidence or history of bleeding diathesis; any hemorrhage or bleeding event CTCAE Grade ≥ 3 or higher within 4 weeks of start of investigational treatment.
* Dehydration CTCAE Grade ≥1
* Unresolved toxicity higher than NCI-CTCAE version 4.0 Grade 1 (excluding alopecia, anemia or lymphopenia) attributed to any prior systemic or radiation therapy or other medical or surgical procedure
* Known hypersensitivity to regorafenib, study drug class, or excipients in the formulation.
* Ongoing or active infection (bacterial, fungal or viral, e.g. human immunodeficiency virus (HIV)) of NCI-CTCAE version 4.0 Grade ≥ 2
* Seizure disorder requiring anti-convulsant therapy (such as steroids or anti-epileptics)
* Pregnancy and lactation (breastfeeding)
* During the study, no other anticancer treatment, including any investigational new drugs, is allowed. Anticancer therapy is defined as any agent or combination of agents with clinically proven anticancer activity. Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy and hormonal therapy during this trial or within 28 days or 5 drug half lives (if drug half-life in subject is known), whichever is shorter (or within 6 weeks or mitomycin C) before start of the study treatment
* Use of hematopoietic growth factors, such as G-CSF (granulocyte colony-stimulating factor), GM-CSF (granulocyte-macrophage colony-stimulating factor), erythropoietin, and interleukin (IL-2, IL-3), within 3 weeks prior to first dose. Subjects taking chronic erythropoietin consistent with institutional guidelines can be included.
* Close affiliation with the investigational site; e.g. a close relative of the investigator or a dependent person (e.g. employee or student of the investigational site)
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
* Inability to swallow oral medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03 (Estimated); Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Peak plasma concentration of regorafenib | 5 days
  Peak plasma concentrations of regorafenib, M-2 and M-5 after single-dose and multiple-dose administration. The outcome will be measured during cycles 1 and 2 using pharmacokinetic blood samples collected on

SECONDARY OUTCOMES:
The area under the concentration-time curve (AUC) for regorafenib | 5 days
  The outcome will be measured during cycles 1 and 2 using pharmacokinetic blood samples collected on days 1, 2, 3 and 5 of both cycles

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sawyer, MD, Principal Investigator — Cross Cancer Institute, Alberta Health Services
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada